CLINICAL TRIAL: NCT02882841
Title: MOlecular BIomarkers and Adherent and Invasive Escherichia Coli (AIEC) Detection Study In Crohn's Disease Patients (MOBIDIC)
Brief Title: MOlecular BIomarkers and Adherent and Invasive Escherichia Coli (AIEC) Detection Study In Crohn's Disease Patients
Acronym: MOBIDIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Enterome (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IBD210
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-04

CONDITIONS: Crohn's Disease
Keywords: AIEC (Adherent and Invasive Escherichia Coli); Mucosal Healing; Non-invasive biomarkers
MeSH Terms: conditions — Crohn Disease | interventions — Biopsy; Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single-arm study (Other)
  Interventions: Other: Biopsies, stool and blood collection

INTERVENTIONS:
Other: Biopsies, stool and blood collection

SUMMARY:
The study is a multicenter, international descriptive study with a bio-collection in 300 evaluable Crohn's disease patients to be processed after usual biological tests via bioinformatics tools.

At this time, this study has no impact neither on treatment nor on disease diagnostic, these will be based on usual medical practices and is no investigational product associated with the conduct of this study.

DETAILED DESCRIPTION:
350 Crohn's disease patients will be included in the study, targeting 300 evaluable patients. An interim analysis will be performed after 50% of the evaluable patients are recruited.

The primary objective is to evaluate the relation between non-invasive biomarkers (host immunological variables and metagenomic analysis in stools) and AIEC detection in biopsies taken during an endoscopy, in order to develop a predictive algorithm of AIEC carriage.

The secondary objectives are:

* Validation of the AIEC detection algorithm using qPCR technology.
* Assessment of the correlation between the presence of AIEC and the endoscopic and clinical evaluations of the disease (CDEIS, SES-CD, Harvey-Bradshaw Index and Crohn's Disease Activity Index).
* Development and validation of a non-invasive qPCR based diagnostic of Mucosal Healing in CD patients.
* Collection of biological samples associated with all clinical and biological data from CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age, inclusive;
* With a diagnosis of ileal or ileo-colonic Crohn's disease for a minimum of 3 months prior to inclusion;
* An ileocolonoscopy scheduled prior to study inclusion;
* Agreeing to participate and to sign an informed consent form;
* Able to perform stool collection, at home, according to protocol;
* Covered by Health Insurance System and/or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

* Colonic Crohn's disease of L2 phenotype based on Montreal classification;
* Extensive small bowel resection (> 100 cm) or short bowel syndrome
* Bowel strictures/stenosis contraindicating ilecolonoscopy;
* Currently with an ostomy or an ileoanal pouch;
* Currently receiving total parenteral nutrition;
* Bowel preparation received in the previous 3 months;
* An increased risk of hemorrhage (patients with anticoagulant/antiplatelet therapy)
* History of intestinal carcinoma and colorectal cancer;
* History or presence of alcohol or substance abuse;
* History of chronic uncontrolled disorders;
* Current participation in an investigational product trial;
* Less than 4 weeks since last participation in a clinical trial;
* Subject inapt or unwilling to participate to the study;
* Pregnant or breastfeeding mother;
* Patient under guardianship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The primary evaluation criterion is the correlation between the detection of AIEC using a non-invasive stool based algorithm and the detection of AIEC using an ileal biopsy taken during an endoscopy. | 6-12 months between inclusion and analysis

CONTACTS AND LOCATIONS:
Locations (3):
- Children's Hospital Boston, Boston, Massachusetts, United States
- Hôpital Saint-Antoine, Paris, France
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No